CLINICAL TRIAL: NCT04188483
Title: Effect of Selenium Supplementation on Immunity Responses to Influenza Vaccination
Brief Title: Effect of Selenium Supplementation on Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery, Deputy Dean of The Second Clinical Medical School,Deputy Dean of Tongji Hospital, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ENT-SELENIUM-01
Record Dates: First submitted 2019-10-13; First posted 2019-12-06 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Selenium Supplementation; Influenza Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selenium Supplementation (Experimental): The selenium supplementation group will receive 200 μg selenium daily by taking two selenium-enriched yeast tablets (SelenoPrecise®, Pharma Nord) once daily for 60 days. Thirty days after the start of the supplementation, the subjects will receive standard seasonal influenza vaccination for the 2019-2020 season.
  Interventions: Dietary Supplement: Selenium Supplementation; Biological: Influenza vaccination
- Non-Selenium Supplementation (Other): The control group will not receive selenium supplementation. Thirty days after allocation, the subjects will receive standard seasonal influenza vaccination for the 2019-2020 season.
  Interventions: Biological: Influenza vaccination

INTERVENTIONS:
Dietary Supplement: Selenium Supplementation — The selenium supplementation group will receive 200 μg selenium daily by taking two selenium-enriched yeast tablets (SelenoPrecise®, Pharma Nord) once daily for 60 days.
  Arms: Selenium Supplementation
Biological: Influenza vaccination — Subjects will receive standard seasonal influenza vaccination for the 2019-2020 season.

SUMMARY:
The study is designed to assess whether selenium supplementation can boost the immunity response to influenza vaccination in healthy adults. This is a randomized, prospective study enrolling a total of 60 healthy subjects, 18-55 years old.

DETAILED DESCRIPTION:
Background: Selenium is an essential trace element required for human health and wellbeing. Despite mouse studies and human clinical trial suggest selenium supplementation might enhance immunity, little is known for the effects of selenium supplementation on humoral immunity. Vaccination is the most effective medical intervention to prevent infections and to reduce disability and mortality associated with infectious disease. However, some individuals, in healthy or disease conditions, mount less effective humoral immune responses to vaccination. Therefore, new strategy to enhance humoral immunity upon vaccination is highly sought after. Using mouse models, we have observed that selenium supplementation significantly increased antigen-specific antibody responses. Thus, we hypothesize that selenium supplementation may be beneficial in enhancing humoral immunity in humans.

Objectives: To investigate whether selenium supplementation will boost the humoral response to influenza vaccination in healthy adults.

Design and trial size: This is a randomized prospective study. A total of 60 healthy subjects, 18-55 years old, will be enrolled in this study.

Intervention and duration: The enrolled subjects will be randomized into selenium supplementation and control group. The selenium supplementation group will receive 200 μg selenium daily by taking two selenium-enriched yeast tablets (SelenoPrecise®, Pharma Nord) once daily for 60 days. The control group will not receive selenium supplementation. Thirty days after allocation, both groups will receive standard seasonal influenza vaccination for the 2019-2020 season. Peripheral blood samples will be collected at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination).

ELIGIBILITY:
Inclusion Criteria:

18-55 years, healthy subjects

Exclusion Criteria:

1. With the history of selenium supplementation as taking supplementation products or living more than 2 years in selenium-enriched area;
2. Had the symptoms of selenium toxicity or serum selenium level greater than 328 μg/L;
3. With the history of the administration of influenza vaccine in past three years or allergic to influenza vaccine;
4. With any current immunologic disorders, including autoimmune and allergic diseases;
5. With any cardiovascular, metabolic, mental, or psychological disorders;
6. Pregnancy or breastfeeding;
7. With the history of infectious diseases including airway infections in past three months;
8. Who are currently participating in other clinical studies or who have participated in other clinical research within 90 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The production of antigen-specific antibodies after vaccination | 60 days
  Viral strain-specific antibodies in serum at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by hemagglutination inhibition (HAI) assay

SECONDARY OUTCOMES:
Immune cell responses after selenium supplementation and vaccination | 60 days
  Frequencies (%) of immune cells including T cells, B cells, monocytes, dendritic cells, NK cells in peripheral blood at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination)will be measured by flow cytometry.
Immune cytokine IFN-γ after selenium supplementation and vaccination | 60 days
  Levels of IFN-γ in plasma at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by enzyme-linked immunosorbent assay (ELISA).
Immune cytokine IL-4 after selenium supplementation and vaccination | 60 days
  Levels of IL-4 in plasma at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by enzyme-linked immunosorbent assay (ELISA).
Immune cytokine IL-10 after selenium supplementation and vaccination | 60 days
  Levels of IL-10 in plasma at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by enzyme-linked immunosorbent assay (ELISA).
Immune cytokine IL-17A after selenium supplementation and vaccination | 60 days
  Levels of IL-17A in plasma at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by enzyme-linked immunosorbent assay (ELISA).
Immune cytokine IL-21 after selenium supplementation and vaccination | 60 days
  Levels of IL-21 in plasma at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by enzyme-linked immunosorbent assay (ELISA).
Selenium levels after selenium supplementation and vaccination | 60 days
  Level of selenium in plasma at baseline (day 0, prior to treatment), day 30, day 37 (7 days after vaccination) and day 60 (30 days after vaccination) will be measured by inductively coupled plasma mass spectrometry (ICP-MS).

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Doctor, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China